CLINICAL TRIAL: NCT04627480
Title: Evaluation of a Neurostimulation Device for Insomnia: A Randomized Trial
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Fisher Wallace (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2513
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-11

CONDITIONS: Insomnia; Insomnia Chronic; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sham Device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experiment Arm (Experimental): Active Fisher Wallace device for full 8 weeks
  Interventions: Device: Fisher Wallace Neurostimulation Device
- Sham Arm (Sham Comparator): Sham Fisher Wallace device for 4 weeks, then cross over at 4 weeks to active device.
  Interventions: Device: Fisher Wallace Neurostimulation Device

INTERVENTIONS:
Device: Fisher Wallace Neurostimulation Device — a Cranial Electrotherapy Stimulator Device (CES).

SUMMARY:
Examine the safety and effectiveness of the Fisher Wallace Cranial Electrotherapy Stimulator Device (CES) for the treatment of insomnia characterized by difficulties with sleep maintenance using a 20-minute treatment right before bedtime.

ELIGIBILITY:
Age greater than or equal to 21 US resident Can receive packages to their home via UPS/Fedex/USPS Read/write English Insomnia Severity Index Score Greater than 14 Diagnosis of insomnia by a medical physician Subjects with a Generalized Anxiety Diagnosis will be excluded Have not contemplated suicide in the past year Not been institutionalized for mental health issues. Not currently being treated for or suspect a mental health issue Not currently experiencing problems with alcohol or drug abuse Can commit to not drinking alcohol 4 hours before bedtime for the duration of the study Not taking medications affecting the nervous system (e.g. psychiatric medications) Not taking hypnotics or any sleep aid or marijuana (in any form) Can commit to one (1) 20 minute session per day for 8 weeks Has not used a brain stimulation treatment in one year No suspected or known history of heart disease No pacemaker, or any form of medical electronics, including but not limited to a deep brain stimulator, electronic stent, etc.

Not under medical supervision for other serious medical condition Not taking opioids No pain or headaches that interrupt sleep Not participating in any other sleep study Not experiencing restless leg syndrome No Nickel Allergy No Sleep Apena as measured by STOP-Bang Assessment

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in total sleep per night at week 4 between active and sham arm | baseline versus week 4
  Measured by Fitbit Charge 4 connected health device work on the wrist

SECONDARY OUTCOMES:
Device Tolerance and Safety measured by SAFTEE | 4 weeks from baseline
  assessment of safety and adverse events
Change in WASO (wake after sleep onset) between sham versus active arms | baseline versus week 4
  measured by Fitbit Charge 4 connected health device worn on the wrist
Change in Insomnia Severity between Sham versus active arms | baseline versus week 4
  measured by the self report Insomnia Severity Index (ISI)

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Remote Virtual Trial), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No